CLINICAL TRIAL: NCT02614469
Title: A Phase 1, Open-label, Randomized, Two-period, Two-treatment, Crossover Study to Evaluate the Effects of Food on the Pharmacokinetics of Urate After a Single Dose of Inosine in Healthy Male Subjects
Brief Title: A Food-Drug Interaction Study of Serum Urate After Oral Inosine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Alan Schwarzschild (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); The Parkinson Alliance (Other)
Responsible Party: Sponsor-Investigator, Michael Alan Schwarzschild, Director, Molecular Neurobiology Laboratory, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INO-PD-P3-2015-FE
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Healthy
MeSH Terms: interventions — Inosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1, Inosine with Food (Experimental): Group 1 subjects will take inosine with food on day 1 after an overnight fast and will take a second dose of inosine without food on day 8 after an overnight fast.
  Interventions: Drug: Inosine
- Group 2, Inosine without Food (Experimental): Group 2 subjects will take inosine without food on day 1 after an overnight fast and will take a second dose of inosine with food on day 8 after an overnight fast.
  Interventions: Drug: Inosine

INTERVENTIONS:
Drug: Inosine — Inosine, 1000 mg

SUMMARY:
The purpose of this study is to assess the effects of food on the amount of urate in the body after a single oral dose of inosine.

DETAILED DESCRIPTION:
Eighteen (18) eligible healthy male subjects will be randomly assigned to two groups with 9 subjects per group to receive a single oral dose of 1000 mg inosine with or without food on day 1 after an overnight fast. Subjects who receive inosine with food on day 1 will receive a second dose of inosine without food on day 8 after an overnight fast. Subjects who receive inosine without food on day 1 after an overnight fast will receive a second dose of inosine with food on day 8 after an overnight fast.

Subjects will be admitted to the clinic before dinner on days 0 and 7, the days before dosing, and will stay in the clinic for 48-h post-dose. During the clinic stay, blood samples will be taken for urate measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 18 and 65 years
2. Body-mass index between 18.0 kg/m2 and 32.0 kg/m2
3. If not surgically sterile, willing to refrain from donating sperm and willing to use appropriate birth control when engaging in sexual intercourse for a period of 90 days following the last dose of the study medication
4. Serum urate < 6.1 mg/dL (approximately 360 μM) at screening
5. Non-smokers for at least 6 months prior to screening
6. Adequate venous access at multiple sites in both arms

Exclusion Criteria:

1. History of alcohol or drug dependence in the past 2 years
2. Had 400 mL of whole blood collection within four months or 200 mL of whole blood collection or who had blood component collection within one month of the screening test
3. Used prescription or over-the-counter (OTC) drugs within 14 days prior to screening
4. Used vitamin preparations or supplements (including St. John's Wort and ginseng) within 28 days prior to the screening test
5. Not willing to refrain from alcohol, grapefruit, grapefruit juice or related products, caffeine consumption (including chocolate), and strenuous exercise within 72 h prior to day 1 and through the end of the PK study
6. Treated with an investigational drug within 30 days or 7 half-lives of the investigational drug, whichever is longer, prior to the first dose of study drug
7. Previously received inosine supplement within three months from the screening or subjects who have had any inosine and suffered an adverse reaction due to it
8. Known HIV disease
9. Had a febrile illness within 5 days prior to the first dose of study medication
10. Vaccinated within 30 days prior to the first dose of medication
11. Has gout or a history or suspicion of kidney stones
12. Determined by the investigator or sub-investigator to be unsuitable for participating in the study based on medical conditions

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason Freeman, M.D., Study Director — Massachusetts General Hospital
Locations (1):
- Covance Clinical Research Unit Inc., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anton FM, Garcia Puig J, Ramos T, Gonzalez P, Ordas J. Sex differences in uric acid metabolism in adults: evidence for a lack of influence of estradiol-17 beta (E2) on the renal handling of urate. Metabolism. 1986 Apr;35(4):343-8. doi: 10.1016/0026-0495(86)90152-6. PMID 3959904
- [Background] Cuhadar S, Koseoglu M, Atay A, Dirican A. The effect of storage time and freeze-thaw cycles on the stability of serum samples. Biochem Med (Zagreb). 2013;23(1):70-7. doi: 10.11613/bm.2013.009. PMID 23457767
- [Background] Dirar AM, A.D., Abdelsalam KEA. Effect of Storage Time and Temperature on some Serum Analytes. International Journal of Pathology 8: 68-71, 2010.
- [Background] Parkinson Study Group SURE-PD Investigators; Schwarzschild MA, Ascherio A, Beal MF, Cudkowicz ME, Curhan GC, Hare JM, Hooper DC, Kieburtz KD, Macklin EA, Oakes D, Rudolph A, Shoulson I, Tennis MK, Espay AJ, Gartner M, Hung A, Bwala G, Lenehan R, Encarnacion E, Ainslie M, Castillo R, Togasaki D, Barles G, Friedman JH, Niles L, Carter JH, Murray M, Goetz CG, Jaglin J, Ahmed A, Russell DS, Cotto C, Goudreau JL, Russell D, Parashos SA, Ede P, Saint-Hilaire MH, Thomas CA, James R, Stacy MA, Johnson J, Gauger L, Antonelle de Marcaida J, Thurlow S, Isaacson SH, Carvajal L, Rao J, Cook M, Hope-Porche C, McClurg L, Grasso DL, Logan R, Orme C, Ross T, Brocht AF, Constantinescu R, Sharma S, Venuto C, Weber J, Eaton K. Inosine to increase serum and cerebrospinal fluid urate in Parkinson disease: a randomized clinical trial. JAMA Neurol. 2014 Feb;71(2):141-50. doi: 10.1001/jamaneurol.2013.5528. PMID 24366103
- [Background] Spitsin S, Hooper DC, Leist T, Streletz LJ, Mikheeva T, Koprowskil H. Inactivation of peroxynitrite in multiple sclerosis patients after oral administration of inosine may suggest possible approaches to therapy of the disease. Mult Scler. 2001 Oct;7(5):313-9. doi: 10.1177/135245850100700507. PMID 11724447
- [Background] Yamamoto T, Moriwaki Y, Cheng J, Takahashi S, Tsutsumi Z, Ka T, Hada T. Effect of inosine on the plasma concentration of uridine and purine bases. Metabolism. 2002 Apr;51(4):438-42. doi: 10.1053/meta.2002.31322. PMID 11912550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects took part in the study at one investigative site in the United States from 15 March 2016 to 10 April 2016.
Groups:
- Group 1, Inosine With Food Then Without Food: Group 1 subjects will take inosine with food on day 1 after an overnight fast and after a 7 day washout, will take a second dose of inosine without food on day 8 after an overnight fast.
  Inosine: Inosine, 1000 mg
- Group 2, Inosine Without Food Then With Food: Group 2 subjects will take inosine without food on day 1 after an overnight fast and after a 7 day washout, will take a second dose of inosine with food on day 8 after an overnight fast.
  Inosine: Inosine, 1000 mg
Period: Period 1
Arm/Group | Group 1, Inosine With Food Then Without Food | Group 2, Inosine Without Food Then With Food
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Group 1, Inosine With Food Then Without Food | Group 2, Inosine Without Food Then With Food
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1, Inosine With Food Then Without Food: Group 1 subjects will take inosine with food on day 1 after an overnight fast and will take a second dose of inosine without food on day 8 after an overnight fast.
  Inosine: Inosine, 1000 mg
- Group 2, Inosine Without Food Then With Food: Group 2 subjects will take inosine without food on day 1 after an overnight fast and will take a second dose of inosine with food on day 8 after an overnight fast.
  Inosine: Inosine, 1000 mg
- Total: Total of all reporting groups
Arm/Group | Group 1, Inosine With Food Then Without Food | Group 2, Inosine Without Food Then With Food | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.44 (16.37) | 34.67 (5.92) | 38.06 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White | 5 | 4 | 9
  Black or African American | 4 | 4 | 8
  Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Maximum Observed Serum Urate Concentration
Time Frame: -12 to 0 hrs pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36 and 48 hrs post-dose
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Inosine Fed: Inosine, 1000 mg tablet, in fed condition, orally once on Day 1 in Period 1 or Day 8 in Period 2.
- Inosine Fasted: Inosine, 1000 mg tablet, in fasted condition, orally once on Day 1 in Period 1 or Day 8 in Period 2.
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 18 | 18
mg/dL | 6.6 (0.7) | 6.4 (0.6)
Statistical Analysis 1: Comparison: Inosine Fed vs Inosine Fasted; To assess the effect of food on the PK of urate, analyses of variance (ANOVA) using a linear mixed-effects model was fitted to the natural logarithmic transformation of PK parameters of urate. The linear mixed-effects model will include subject as a random effect, and treatment, period, and sequence as fixed effects. The 90% confidence intervals were constructed for the ratio of geometric means of PK parameters between fed and fasted treatments, based on log-transformed data; Test type: Superiority or Other; Ratio of Geometric Means = 103, 90% CI 2-sided [98.0 to 108] — Fed/Fasting Ratio

2. Primary Outcome: AUC (0-t): Area Under the Serum Concentration-time Curve From Time 0 to Time t (Time of Last Quantifiable Plasma Concentration)
Time Frame: -12 to 0 hr pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 hrs post-dose
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 18 | 18
mg*hr/dL | 267 (30.2) | 268 (26.4)
Statistical Analysis 1: Comparison: Inosine Fed vs Inosine Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of Geometric Means = 99.3, 90% CI 2-sided [96.9 to 102] — Fed/Fasted Ratio

3. Primary Outcome: AUC (0-inf): Area Under the Serum Concentration-time Curve From Time 0 to Infinity
Time Frame: -12 to 0 hr pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 hrs post-dose
Population: AUC (0-inf) of 1 subject was not able to be calculated based on the serum concentration-time curve of the subject.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 17 | 17
mg*hr/dL | 2040 (2261) | 2031 (2278)

4. Primary Outcome: Tmax: Time of Maximum Serum Concentration
Time Frame: -12 to 0 hr pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 hrs post-dose
Measure: Median (Full Range); unit: hr
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 18 | 18
hr | 3.0 [1.0 to 6.0] | 3.0 [1.0 to 24.0]

5. Primary Outcome: T1/2: Apparent Terminal Half-life
Time Frame: -12 to 0 pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 hrs post-dose
Population: T 1/2 of 1 subject was not able to be calculated based on the serum concentration-time curve of the subject.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 17 | 17
hr | 242 (341) | 241 (331)

6. Primary Outcome: Baseline Corrected Cmax: Baseline Corrected Maximum Serum Concentration
Description: Correction for individual endogenous urate levels was done by subtracting the individual mean endogenous baseline concentration prior to dosing from each post-dose concentration in the profile. The two samples collected at -12 h and 0 h (pre-dose) before the meal were used to measure the mean endogenous baseline concentrations in each dosing period (periods 1 and 2). Negative concentrations were set to zero.
Time Frame: -12 to 0 hr pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 hrs post-dose
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 18 | 18
mg/dL | 1.73 (0.46) | 1.65 (0.37)
Statistical Analysis 1: Comparison: Inosine Fed vs Inosine Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of Geometric Means = 103, 90% CI 2-sided [90.9 to 118] — Fed/Fasted Ratio

7. Primary Outcome: Baseline Corrected AUC (0-t): Baseline Corrected Area Under the Serum Concentration-time Curve From Time 0 to Time t (Time of Last Quantifiable Serum Concentration)
Description: as for outcome 6
Time Frame: -12 to 0 hr pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 hrs post-dose
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 18 | 18
mg*hr/dL | 36.1 (15.1) | 39.3 (13.3)
Statistical Analysis 1: Comparison: Inosine Fed vs Inosine Fasted; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of Geometric Means = 83.4, 90% CI 2-sided [62.1 to 112] — Fed/Fasted Ratio

8. Primary Outcome: Baseline Corrected AUC (0-inf): Baseline Corrected Area Under the Serum Concentration-time Curve From Time 0 to Infinity
Description: Correction for individual endogenous urate levels was done by subtracting the individual mean endogenous baseline concentration prior to dosing from each post-dose concentration in the profile. The two samples collected at -12 h and 0 h (pre-dose) before the meal were used to measure the mean endogenous baseline concentrations in each dosing period (periods 1 and 2).
Time Frame: -12 to 0 hr pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, and 48 hrs post-dose
Population: Baseline Corrected AUC (0-inf) values of 2 subjects were not able to be calculated based on the serum concentration-time curve of these subjects.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 16 | 16
mg*hr/dL | 80.4 (84.2) | 83.0 (86.3)

9. Primary Outcome: Baseline Corrected Tmax: Baseline Corrected Time of Maximum Serum Concentration
Description: as for outcome 8
Time Frame: -12 to 0 h pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, and 48 hrs post-dose
Measure: Median (Full Range); unit: hr
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 18 | 18
hr | 3.0 [1.0 to 6.0] | 3.0 [1.0 to 24.0]

10. Primary Outcome: Baseline Corrected T1/2: Baseline Corrected Apparent Terminal Half-life
Description: as for outcome 8
Time Frame: -12 to 0 hr pre-dose and 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 36, 48 hrs post-dose
Population: Baseline Corrected T 1/2 values for 2 subjects were not able to be calculated based on the serum concentration-time curve of these subjects.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 16 | 16
hr | 44.3 (71.5) | 44.7 (76.2)

11. Secondary Outcome: Safety Assessment (Vital Signs)
Description: Number of participants with clinically significant findings in vital signs by investigator after study drug administration.
Time Frame: Up to 10 days after first study drug administration at Day 1 of Period 1
Measure: Number; unit: participants
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 18 | 18
participants | 0 | 0

12. Secondary Outcome: Safety Assessment: Adverse Events
Description: Number of participants with adverse events after study drug administration
Time Frame: Up to 10 days after first study drug administration at Day 1 of Period 1
Measure: Number; unit: participants
Arm/Group | Inosine Fed | Inosine Fasted
Number analyzed (Participants) | 18 | 18
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 9 days after first dosing at Day 1 of Period 1, or Day 10 of Period 2
Arm/Group | Inosine Fed | Inosine Fasted
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data and results and all intellectual-property rights in the data and results derived from the study will be the property of the sponsor. No publication or disclosure of study results will be permitted except as specified in a separate, written agreement between the Sponsor and the Investigator. If results of this study are reported in medical journals or at meetings, all subjects' identities will remain confidential.